CLINICAL TRIAL: NCT02305069
Title: The Effect of Obesity-induced Cytokine Elevation on the Molecular Regulation of Protein Turnover and Carbohydrate Metabolism in Human Skeletal Muscle
Brief Title: Effect of Obesity-derived Cytokines on Protein Turnover and Carbohydrate Metabolism in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RIS33323
Record Dates: First submitted 2014-11-10; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Obesity; Sarcopenia
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Pioglitazone; Insulin; Octreotide; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet taken once daily for 12 weeks.
  For study visits performed pre- and post 12-week placebo treatment for the assessment of muscle protein synthesis and leg protein breakdown, the following substances are administered as part of the analytical technique: insulin, octreotide, glucose, mixed amino acids, [2H5]phenylalanine and [1-13C]leucine. The doses administered change as the analytical technique is conducted and for clarity are described in detail in the protocol.
  Interventions: Drug: Insulin; Drug: Octreotide; Drug: Glucose; Drug: Mixed Amino Acids; Other: [2H5]phenylalanine; Other: [1-13C]leucine
- Pioglitazone (Experimental): 30mg pioglitazone encapsulated and taken once daily for 12 weeks.
  For study visits performed pre- and post 12-week pioglitazone treatment for the assessment of muscle protein synthesis and leg protein breakdown, the following substances are administered as part of the analytical technique: insulin, octreotide, glucose, mixed amino acids, [2H5]phenylalanine and [1-13C]leucine. The doses administered change as the analytical technique is conducted and for clarity are described in detail in the protocol.
  Interventions: Drug: Pioglitazone; Drug: Insulin; Drug: Octreotide; Drug: Glucose; Drug: Mixed Amino Acids; Other: [2H5]phenylalanine; Other: [1-13C]leucine

INTERVENTIONS:
Drug: Pioglitazone — Described elsewhere
  Other Names: Actos
  Arms: Pioglitazone
Drug: Insulin — Administered to simulate the feeding response in study visits. Description of amount administered provided elsewhere.
  Other Names: Actrapid
Drug: Octreotide — Administered to simulate the feeding response in study visits. Description of amount administered provided elsewhere.
  Other Names: Sandostatin
Drug: Glucose — Administered to simulate the feeding response in study visits. Description of amount administered provided elsewhere.
  Other Names: Dextrose
Drug: Mixed Amino Acids — Administered to simulate the feeding response in study visits. Description of amount administered provided elsewhere.
  Other Names: Glamin
Other: [2H5]phenylalanine — Administered to allow the determination of leg protein breakdown rates in study visits. Description of amount administered provided elsewhere.
Other: [1-13C]leucine — Administered to allow the determination of muscle protein synthesis rates in study visits. Description of amount administered provided elsewhere.

SUMMARY:
Obesity in humans has been shown to result in the increased release of small inflammatory-inducing proteins, called cytokines, from the fat cells of the body. The investigators are interested in the effects of these cytokines on the mechanisms that control muscle mass and metabolism in the obese human. Previous research from work in cells and animals has shown the cytokines reduce the synthesis of muscle proteins and simultaneously enhance their rate of breakdown, resulting in a loss of muscle mass. Furthermore, research suggests that the same cytokines may inhibit carbohydrate oxidation, a pivotal step in muscle metabolism. However, despite these potential negative consequences for skeletal muscle function, the effect of low-level and persistent inflammation as seen in obese humans, remains largely unknown.

In the current study, the investigators plan to measure the rates of synthesis and breakdown of muscle proteins in conjunction with rates of carbohydrate oxidation in obese older participants, and compare them to rates determined in healthy non-obese individuals. Furthermore, participants will undergo a 12-week course of either pioglitazone, an insulin sensitiser often prescribed to type II diabetics, or a placebo. Pioglitazone has been shown previously to normalise the levels of cytokines in the blood of chronically inflamed individuals. By repeating after the 12-week intervention period the initial measurements described above, and by accurately determining the levels of the cytokines, the identification of the negative effects of obesity-induced inflammation in older adults on muscle metabolism will be determined.

DETAILED DESCRIPTION:
Recruitment of subjects:

24 obese (but otherwise healthy) participants with elevated cytokine levels and 24 non-obese subjects with normal cytokine levels will be recruited. Following the first experimental visit (see below), participants will be divided in a double-blind fashion into four groups (n=12). In previous studies utilising similar low-grade inflammatory states where thiazolidinediones have been administered, significant differences (P<0.05) in processes under investigation have been observed with group sizes of 10. Therefore group sizes of 12 have been selected to accommodate for the anticipated 15% dropout seen in long-term studies. Participants will be male, age matched (>55 years), non-smoking, live a sedentary lifestyle and non-vegetarian. Before taking part in the study, all subjects will undergo medical screening and complete a general health questionnaire. This will include measures of blood pressure, heart rate, 12-lead electrocardiogram (ECG), blood biochemistry and a blood clotting profile. For non-control subjects, inclusion into the study will be determined by measures of waist circumference (>100 cm), and inflammatory status (non-obese subjects with C-reactive proteins (CRP) plasma levels <1.35 μg.ml-1 and tumor necrosis factor-alpha (TNFα) plasma levels <3.3 pg.ml-1 and obese subjects with a CRP >1.35 μg.ml-1 and TNFα >4.1 pg.ml-1). Following an explanation of the study and associated procedures, written consent will be obtained and subjects made aware that they are free to withdraw at any point. Subjects will be recruited via press advertisements from the local population.

Experimental trials:

At the start of a 12-week long study, muscle protein synthesis and leg protein breakdown will be determined in all subjects via the administration of stable-isotopes of leucine and phenylalanine concomitant to a two-stage insulin clamp to simulate going from the fasted to fed state. This will establish the baseline values for these measures prior to the 12-week intervention period. These measures will be achieved in a single visit with the execution of an established protocol for the determination of muscle protein synthesis and leg protein breakdown. In summary, to achieve this the following will be performed: a basal muscle biopsy from the thigh will be obtained after which serum insulin concentrations will be held at fasting levels and a further muscle biopsy obtained; once taken serum insulin concentrations will be elevated and mixed amino acids administered to simulate feeding followed by the taking of a third and final muscle biopsy. The taking of biopsies will allow for the determination of isotope incorporation and thereby the determination of muscle protein synthesis and leg protein breakdown rates.

Following the first experimental visit, subjects will start a 12 week treatment period of either pioglitazone (30 mg•day-1) or a placebo, administered in a double-blind fashion. Subjects will be monitored at intervals throughout the period to ensure compliance and report unwanted side effects. After 12 weeks of drug or placebo administration, subjects will return to the laboratory for a repeat of the measurements determined in the first experimental visit (muscle protein synthesis and leg protein breakdown in response to simulated feeding). Circulating levels of select cytokines will be additionally examined in blood samples collected from subjects at the start of the two experimental visits (pre- and post- 12-week drug intervention period), thus allowing an assessment of any associated changes between systemic cytokine concentrations and muscle protein synthesis and leg protein breakdown.

Study protocol:

The study involves two visits separated by a 12-week drug intervention period. At each of the two visits muscle protein synthesis and leg protein breakdown rates in response to simulated feeding are to be assessed using an established experimental protocol described below:

Subjects will be asked to abstain from alcohol and exercise for 48 h prior to each experimental visit and to arrive on the morning of the experimental visit in a fasted state. Subjects will be asked to rest in a semi-supine position while a cannula is inserted retrograde into a superficial vein on the dorsal surface of the non-dominant hand for blood sampling. The hand will be kept in a hand-warming unit (air temperature 50-55°C) to arterialise the venous drainage of the hand. A cannula will be placed in an antecubital vein in each forearm for the infusion of insulin, octreotide, glucose, amino acids and stable-isotope infusions of leucine and phenylalanine to simulate feeding in precise manner; a catheter placed in the femoral vein will allow, in conjunction with arterialised-venous (A-V) blood samples, arterial and venous blood sampling across the leg. To assess muscle protein synthesis and leg protein breakdown rates in response to feeding, serum insulin will initially be maintained at fasting concentrations by the administration of insulin (0.6 mU•m-2•min-1) for 120 minutes and, to prevent endogenous insulin production, Octreotide (30 ng•kg-1•min-1). Then, to simulate feeding, serum insulin concentrations will be increased equivalent to the fed state for 120 minutes (~40 mU•l-1) and 20g of mixed amino acids (Glamin® Fresenius-Kabi, UK) administered by infusion in conjunction with glucose to stabilise blood glucose concentrations (~4.5 mmol.l-1). Infusions of stable isotope versions of phenylalanine and leucine will be maintained throughout the experimental visit. Initially, a single priming dose of [2H5]phenylalanine (0.33 mg•kg-1 body mass, 98 atom % excess) and [1-13C]leucine (0.8 mg•kg-1 body mass, 99 atom % excess) will be administered, followed by a constant infusion of 0.5 mg•kg-1•h-1 phenylalanine and 1.0 mg•kg-1•h-1 leucine. The use of these two stable-isotopes in combination with muscle biopsies obtained from the vastus lateralis muscle of the leg at t = 0, 120 and 240 min and blood sampling throughout the visit, will allow muscle protein synthesis and leg protein breakdown rates in response to feeding to be calculated. At regular intervals throughout the experimental period, respiratory gas exchange will be monitored by measuring oxygen (O2) uptake and carbon dioxide (CO2) production using a ventilated hood indirect calorimeter (NutrEn, UK) to calculate the respiratory exchange ratio.

After completion of the initial visit where baseline measures of muscle protein synthesis and leg protein breakdown in response to feeding have been established, the 12-week drug intervention period will begin. On completion of the 12-week intervention, the study visit described above will be repeated to determine the effects of the intervention on the outcome measures listed.

Sample collection:

At the start of each experimental visit, 8 ml of blood will be collected from a venous cannula into ethylenediaminetetraacetic acid (EDTA) vacutainers. Following centrifugation at 4°C, the extracted plasma will be stored at -80°C to allow the later determination of circulating levels of select cytokines. During the insulin clamp, 1 ml of A-V blood will be obtained every 5 min for the monitoring of blood glucose concentration (YSI 2300 STATplus, Yellow Springs Instruments, USA). A-V blood (5 ml) will be collected at baseline and at +30, +75, +90, +105, +120, +150, +195, +210, +225, +240 min, allowed to clot, centrifuged, and the serum stored in liquid nitrogen. Insulin will be measured in these samples at a later date with a radioimmunoassay kit (Coat-a-Count Insulin, USA). Femoral venous and A-V blood samples (2 ml) will be taken for blood tracer measurements at -5, +75, +90, +105, +120, +195, +210, +225, +240 min, centrifuged at 4°C and stored at -80°C. Muscle biopsies will be obtained from the vastus lateralis muscle at 0, +120 and +240 min using the percutaneous needle biopsy technique. Muscle samples will be snap frozen in liquid nitrogen prior to the determination of [1-13C]leucine incorporation.

After-care of the subjects:

Auditing of the Investigator's past studies involving muscle biopsies and cannulation procedures has shown the procedures to be well tolerated by subjects and to have few significant complications. Scarring of the skin is minimal and invisible after a few months. All muscle biopsies are obtained under sterile conditions by medically qualified staff and after the injection of local anaesthetic. All subjects are carefully monitored before, during, and after the procedure to ensure that they are comfortable at all times. After each biopsy, the skin is closed with a sterile adhesive strip and covered with a waterproof adhesive dressing. On removal of the cannulae, pressure is applied to stop bleeding, and the sites dressed with a waterproof adhesive dressing. Subjects are given a leaflet before they leave the laboratory containing after-care information and contact details of our clinicians should they need advice. Further, subjects will be contacted by telephone on weeks 2, 6 & 10 to confirm the absence of any adverse effects of the drug administration. Subjects will also be provided with contact details that they can use should they have any concerns.

Measurements and analysis:

Muscle biopsy samples and blood samples shall be measured for tracer incorporation, allowing rates of muscle protein synthesis and breakdown to be calculated. Collected blood samples will be analysed for circulating levels of cytokines. By performing these measurements pre- and post- pioglitazone treatment, the consequences of inflammation in aged individuals on muscle metabolism will be determined. Statistical analysis shall be performed using analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Male
* 55-75 years old
* Body Mass Index 20-25 or >30 kg/m2
* Residing in Nottinghamshire area

Exclusion Criteria:

* Taking statin medication
* Clotting disorders of previous central venous access (CVA) / thrombosis-inducing activity (TIA)/ deep vein thrombosis (DVT)
* Metabolic disease e.g. diabetes, thyroid dysfunction
* Inflammatory conditions e.g. Rheumatoid Arthritis, Crohn's Disease
* Tobacco smoker in previous 3 years
* Lower limb circulation problems e.g. Claudication
* Epilepsy
* Renal pathology
* Respiratory problems including asthma

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein synthesis response to simulated feeding with data reported as % fractional synthetic rate per hour. | Assessed at study visits pre and post 90 day drug intervention period

SECONDARY OUTCOMES:
Change in leg protein breakdown response to simulated feeding with data reported as nmol/min/100g leg mass. | Assessed at study visits pre and post 90 day drug intervention period
Change in respiratory exchange ratio response to simulated feeding with data reported as the ratio between the volume of CO2 produced and O2 consumed in air breathed. | Assessed at study visits pre and post 90 day drug intervention period
Change in plasma concentration of pro-inflammatory cytokines with data reported as picograms per ml of plasma. | Assessed pre- and post- 90 day drug intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Greenhaff, PhD, Principal Investigator — The University of Nottingham
Locations (1):
- David Greenfield Physiology Laboratories, Nottingham, Nottinghamshire, United Kingdom